CLINICAL TRIAL: NCT04592731
Title: A Clinical Trial to Evaluate the Efficacy and Safety of Acetylated Natural Nucleotides in Treating Hand-foot Syndrome (HFS)
Brief Title: Acetylated Natural Nucleotides in Treating Hand-foot Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nan xu (Other)
Responsible Party: Sponsor-Investigator, Nan xu, Department Head in Dermatology, Shanghai East Hospital
Organization: Shanghai East Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEH001
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hand-foot Syndrome
MeSH Terms: conditions — Hand-Foot Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gel containing Acetylated Natural Nucleotides (Experimental)
  Interventions: Drug: Gel containing Acetylated Natural Nucleotides
- Vehicle Gel (Placebo Comparator)
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: Gel containing Acetylated Natural Nucleotides — The study drug is a gel containing acetylated natural nucleotides.
  Arms: Gel containing Acetylated Natural Nucleotides
Drug: Vehicle Gel — The vehicle gel contains no acetylated natural nucleotides but with the same base as study drug.
  Arms: Vehicle Gel

SUMMARY:
The clinical trial is planned to investigate the efficacy and safety of acetylated natural nucleotides in treating anti-cancer medications induced hand-foot syndrome (HFS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Pathologically conﬁrmed cancer receiving capecitabine-based anti-cancer therapy (capecitabine with or without other anti-cancer drugs).
* With HFS determined by "CTCAE v5.0 - PPE" as grade 2 or above.
* Able to use topical medications and complete questionnaires reliably with or without assistance.
* ECOG performance score < 2.

Exclusion Criteria:

* Has HFS due to other medications and does not recover within 4 weeks prior to baseline.
* Other skin disorders that will affect efficacy evaluation on the hands and feet, including but not limited to: tinea of feet and hands, hand/foot eczema, palmoplantar pustulosis, palmoplantar keratosis, acrodermatitis continua etc.
* Uncontrolled intercurrent illness as determined by the investigator including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, recent myocardial infarction, uncontrolled hypotension or hypertension, cardiac arrhythmia, or psychiatric illness and social situations that would limit compliance with study requirements.
* Significantly abnormal lab test:

  * Inadequate hematologic function as indicated by:

    * Absolute neutrophil counts (ANC) < 1,500 /mm^3
    * Hemoglobin (Hgb) < 8.5 g/dL
    * Platelet count < 75,000 /mm^3
    * PT or PTT > 1.5 x ULN (if patients on anticoagulants: PT INR > 3.5 x ULN)
  * Inadequate renal and liver function as indicated by:

    * Albumin < 2.8 g/dL
    * Total bilirubin > 1.5 x ULN (or > 2.5 x ULN for patients with Gilbert's syndrome)
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase > 2 x ULN
    * Creatinine > 2 x ULN
* Any other condition which, in the opinion of the Investigator, would impede compliance, hinder completion of the study, compromise the well-being of the patient, or interfere with the study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve "NCI CTCAE v5.0 - Palmar-Plantar Erythrodysesthesia (PPE)" grade 0 or 1 | 6 weeks
  The proportion of patients who achieve "NCI CTCAE v5.0 - PPE" grade 0 or 1 at week 6 from grade 2 or above at baseline

SECONDARY OUTCOMES:
Safety of study drug | 6 weeks
  Safety of study drug as determined by number of participants with abnormal laboratory values and/or Adverse Events that are related to treatment
Proportion of patients who achieve at least one grade improvement in HFS severity | 6 weeks
  The proportion of patients who achieve at least one grade improvement in HFS severity according to "NCI CTCAE v5.0 - PPE" by week 6
Change from baseline in patient reported pain using Visual Analog Scale (VAS) | 6 weeks
  Change from baseline in patient reported pain using VAS at week 6. VAS is a scale used to determine the pain intensity experienced by individuals, which consists of a line 10 cm in length, with the left side signifying no pain and the right side signifying the worst pain ever.
Change from baseline in Hand-Foot Skin Reaction and Quality of Life (HF-QoL) Questionnaire total score | 6 weeks
  Change from baseline in HF-QoL Questionnaire total score at week 6. HF-QoL questionnaire is comprised of a 20-item symptom domain and an 18-item daily activity domain. Each item is rated on a 5-point scale from 0 (not at all) to 4 (always or extremely) during the previous week. The HF-QoL symptom and daily activity total scores are transformed to a scale of 0 to 100, based on the sum of each unit-weighted item score divided by the maximum score. Higher scores on the HF-QoL indicate worse quality of life or greater symptom burden.
The proportion of patients whose anti-cancer medications are impacted due to HFS | 6 weeks
  The proportion of patients who need temporary interruption or permanent discontinuation and/or dose reduction of anti-cancer medications due to HFS

CONTACTS AND LOCATIONS:
Overall Officials: Nan Xu, M.D., Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No